CLINICAL TRIAL: NCT04216628
Title: Early Versus Late Amniotomy Following EAB Cervical Ripening - Does Parity Matter?
Brief Title: Early Versus Late Amniotomy Following EAB Cervical Ripening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to difficulties in recruitment
Sponsor: Assuta Ashdod Hospital (Other)
Collaborators: Wolfson Medical Center (Other Government); Rambam Health Care Campus (Other); The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Eran Brazilay, MD PhD, Senior physician, OBGYN department, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-19-AAA
Record Dates: First submitted 2019-12-11; First posted 2020-01-03 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: Amniotomy; Cervical ripening; Oxytocin; Exrea amniotic baloon
MeSH Terms: interventions — Amniotomy; Oxytocin

STUDY DESIGN:
Intervention Model Description: 1. For the early amniotomy group amniotomy will be performed as the exclusive primary intervention. Oxytocin infusion will begin as per local standard dose protocol no earlier than 2 hours following amniotomy.
  2. For the late amniotomy group oxytocin infusion will begin as per local standard dose protocol. Amniotomy will be performed no earlier than 2 hours following the commence of oxytocin infusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early amniotomy group (Other): Amniotomy will be performed as the exclusive primary intervention. Oxytocin infusion will begin as per local standard dose protocol no earlier than 2 hours following amniotomy.
  Interventions: Other: Amniotomy
- Late amniotomy group (Other): Oxytocin infusion will begin as per local standard dose protocol. Amniotomy will be performed no earlier than 2 hours following the commence of oxytocin infusion
  Interventions: Other: Amniotomy

INTERVENTIONS:
Other: Amniotomy — Artificial rupturing of membranes and IV infusion of Oxytocin
  Other Names: Oxytocin

SUMMARY:
The objective of this study is to investigate the course of labor in early versus late amniotomy following balloon cervical ripening in women undergoing term induction of labor stratified by parity.

DETAILED DESCRIPTION:
Induction of labor is a common obstetric procedure with a reported rate of 23.3% in 2012 in the United State. It has been recently reported that Induction of labor at full term in uncomplicated singleton gestations is not associated with increased risk of cesarean delivery and overall has similar outcomes compared to expectant management.

Induction of labor in women with an unripened cervix is comprised of two stages, cervical ripening followed by augmentation of labor.

Extra amniotic balloon inflation is a widespread mechanical method of cervical ripening that commonly results in a ripened cervix open to 3-4 cm without significant uterine contractions. At this point the clinician may opt to perform artificial rupture of membranes or rather first begin oxytocin infusion delaying amniotomy to later stages of labor. A retrospective cohort showed early amniotomy after Foley balloon catheter removal was associated with shorter duration of labor induction among nulliparous women.In accordance, an RCT investigating the efficacy of early amniotomy in nulliparous women showed this practice resulted in labor shortening without increasing the rate of cesarean section, yet these women were treated by different methods for cervical ripening. Contradicting results were shown in a randomized controlled trial addressing the very question of early versus late amoniotomy after balloon ripening, concluding that postponing amniotomy until active labor commences results in a reduction of dystocia indicated cesarean section. However no distinction was made in this study between nulliparous and multiparous parturients. Since these comprise different groups with distinct labor curves, the question remains whether one should consider parity when deciding to perform early vs late amniotomy following balloon expulsion.

Both Amniotomy and Oxytocine infusion are part of the routine protocol and necessary procedures for induction of labor. Adverse outcome of amniotomy includes fetal heart rate changes, cord prolapse and intrapartum fever when labor is prolonged. Adverse outcome of oxytocine include hypertonus and fetal heart rate changes requiring cessation of oxytocine infusion (as in routine protocol) and intrapartum fever if labor is prolonged (not due to oxytocine infusion per se). Most of the patients admitted for induction of labor will need both amniotomy and oxytocine, however the role of the order of these two procedures is unclear ,as well as whether the order of these procedures affect the rate of adverse outcome.

The objective of this study is to investigate the course of labor in early versus late amniotomy following balloon cervical ripening in women undergoing term induction of labor stratified by parity.

STUDY PROTOCOL Multicenter randomized control trial that will be conducted in 4 medical centers in Israel.

Women with a singleton viable gestation undergoing indicated labor induction at term (37-42 weeks of gestation) who undergoing induction of labor at term with a low bishop score<4 who require extra amniotic balloon cervical ripening will be asked to participate in the study. Written informed consent will be obtained from all patients.

Early amniotomy- Amniotomy performed as the exclusive primary intervention to augment labor following expulsion of the EAB regardless of cervical dilatation.

Late amniotomy- EAB expulsion is followed by oxytocin infusion at increasing increments as the primary intervention as an exclusive intervention for at least 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 37-42 weeks
2. Singleton pregnancy
3. Vertex presentation
4. Medical indication for induction of labor
5. Need for cervical ripening (Bishop score <=6)
6. Consent to participate in the study
7. Women age at or >18 years

Exclusion Criteria:

1. Multiple pregnancies
2. Preterm pregnancy
3. Previous cesarean section
4. Uterine malformation
5. Withdrawal of consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Induction of labor :
  Women with a singleton viable gestation undergoing indicated labor induction at term (37-42 weeks of gestation).
Enrollment: 146 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Time to delivery | Up to 96 Hours
  The time from induction defined as the primary intervention following balloon expulsion to delivery.
Delivery within 24 hours | Up to 96 Hours
  The proportion of women that delivered within 24 hours of induction

SECONDARY OUTCOMES:
Cesarean delivery | Up to 96 Hours
  Cesarean delivery rates and indications
Operative delivery | Up to 96 Hours
  Operative delivery rates and indications
Intrapartum fever | Up to 96 Hours
  Fever >38 degrees Celsius during labor
Postpartum fever during the postpartum hospital stay | Up to 7 days
  Fever >38 degrees Celsius > 24hours after delivery
Post partum hemorrhage | Up to 7 days
  Estimation of obstetrician >500cc bleeding post partum for vaginal delivery or>1000 cc at cesarean section
Neonatal outcomes- Apgar | 10 minutes
  Apgar score
Neonatal outcomes - PH umbilical | 10 minutes
  PH of vein and or artery of umbilical cord
Neonatal outcomes- NICU admission | Up to 30 days
  Admission to Neonatal Intensive Care Unit
Neonatal outcomes- infection | Up to 30 days
  Neonatal fever/sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Yael Ganor Paz, MD, Principal Investigator — Assuta Ashdod medical center
Locations (1):
- Assuta Ashdod, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osterman MJ, Martin JA. Recent declines in induction of labor by gestational age. NCHS Data Brief. 2014 Jun;(155):1-8. PMID 24941926
- [Background] Saccone G, Berghella V. Induction of labor at full term in uncomplicated singleton gestations: a systematic review and metaanalysis of randomized controlled trials. Am J Obstet Gynecol. 2015 Nov;213(5):629-36. doi: 10.1016/j.ajog.2015.04.004. Epub 2015 Apr 13. PMID 25882916
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Macones GA, Cahill A, Stamilio DM, Odibo AO. The efficacy of early amniotomy in nulliparous labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):403.e1-5. doi: 10.1016/j.ajog.2012.08.032. Epub 2012 Aug 24. PMID 22959833
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Schoen CN, Grant G, Berghella V, Hoffman MK, Sciscione A. Intracervical Foley Catheter With and Without Oxytocin for Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jun;129(6):1046-1053. doi: 10.1097/AOG.0000000000002032. PMID 28486381
- [Background] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Background] Levy R, Ferber A, Ben-Arie A, Paz B, Hazan Y, Blickstein I, Hagay ZJ. A randomised comparison of early versus late amniotomy following cervical ripening with a Foley catheter. BJOG. 2002 Feb;109(2):168-72. doi: 10.1111/j.1471-0528.2002.01137.x. PMID 11888099